CLINICAL TRIAL: NCT01619228
Title: Ontogeny of Skin Barrier Maturation in Premature Infants
Brief Title: Skin Maturation in Premature Infants
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: CCHMC IRB 2011-1840
Record Dates: First submitted 2012-06-04; First posted 2012-06-14 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2018-05

CONDITIONS: Premature Birth of Newborn
Keywords: premature infant; neonate; skin maturation; stratum corneum maturation; ontogeny of neonatal skin maturation; sunflower oil; effect of Vitamin B3 on premature skin maturation; skin acidity; stratum corneum barrier integrity; stratum corneum lipid composition; stratum corneum biomarkers; stratum corneum cytokines; stratum corneum structural proteins
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full thickness tissue samples are to be collected from subjects who undergo surgery as part of their care and for whom a sample of tissue can be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Premature Infants: Infants born at < 37 weeks gestational age
- Full Term Infants: Infants born at equal to or greater than 37 weeks gestational age
- Adults: Adults are parents of infants enrolled in the study

SUMMARY:
The skin barrier lipids will be lower in premature infants than in full term infants and will become normal over 3-4 months after birth. The higher skin pH in premature infants will be related to an altered lipid composition which will change as the skin acidifies.

DETAILED DESCRIPTION:
Premature infants have a poor epidermal barrier with few cornified layers, putting them at significant risk for increased permeability to external agents, skin compromise, high water loss and infection. While the skin develops rapidly after birth upon exposure to the dry environment, the ontogeny of the skin maturation and the time to a fully functional and protective stratum corneum (SC) barrier is largely unknown. The impact of a poor skin barrier on nosocomial infections and the morbidity associated with prematurity is not well defined. The purpose is to evaluate skin barrier maturation in premature infants compared to full term infants. The skin barrier lipids will be lower in premature infants than in full term infants and will become normal over 3-4 months after birth. The higher skin surface acidity in premature infants will be related to an altered lipid composition which will change as the skin acidifies.

Full thickness skin samples will be collected from premature and full term infants during the time of medically necessary surgical procedures for genomic/transcriptomics analyses. The gene profiles will be compared to the corresponding biomarker profiles to determine the relationship between genes and gene expression products, i.e., biomarkers. The genomic/transcriptomics, biomarker, instrumental and clinical assessments will be examined for relationships and compared between premature and full term cohorts.

ELIGIBILITY:
Inclusion Criteria:

(1) Premature infants of gestational ages 24 to 36.9 weeks or healthy full term infants of gestational age ≥ 37 weeks (2) Premature infants who are patients in the Neonatal Intensive Care Unit of University Hospital (3) Healthy full term infants (who were born at University Hospital (4) Full term infants (≥ 37 weeks gestational age) who were transported to Cincinnati Children's Hospital Medical Center for care after birth (4) Free of congenital conditions known to affect the skin such as epidermolysis bullosa, ichthyosis, trisomy 2 (5) Free of skin infections such as herpes simplex (6) Sufficiently medically stable such that study procedures can be tolerated (7) Parent/guardian willing to provide written informed consent for participation

Direct admit surgical subjects

Inclusion Criteria:

1. Premature infants of gestational ages 24 to 36.9 weeks
2. Full term infants ≥ 37 weeks gestational age

(2) Infant admitted directly to the Neonatal Intensive Care Unit of Cincinnati Childrens for surgical procedures after delivery (3) Free of congenital conditions known to affect the skin such as epidermolysis bullosa, ichthyosis and trisomy 21 (5) Free of skin infections such as herpes simplex (4) Sufficiently medically stable such that study procedures can be tolerated (5) Parent/guardian willing to provide written informed consent for participation

Exclusion Criteria:

1. Gestational age < 24 weeks
2. Have congenital conditions that affect the skin such as epidermolysis bullosa, ichthyosis, trisomy 21
3. Have a skin infection such as herpes simplex
4. Judged to be medically unstable such that study procedures cannot be tolerated
5. Parent/guardian unwilling to provide written informed consent for participation.

Direct admit surgical subjects

Exclusion Criteria:

1. Infants ≥ 43 weeks gestational age
2. Have congenital conditions known to affect the skin such as epidermolysis bullosa, ichthyosis, trisomy 21
3. Have a skin infection such as herpes simplex

Adult subject controls:

Inclusion Criteria:

1. Parent of an infant enrolled in the study
2. Free from skin irritation, rash, scars, wounds or other skin damage in an area of at least 200 cm2 on one volar forearm
3. Able to come to the infant's hospital for study measurements on one day when infant measurements are made
4. Willing to provide written informed consent for participation

Exclusion Criteria:

(1) Not a parent of an infant enrolled in the study (2) Have skin irritation, rash, scars, wounds or other skin damage in an area of at least 200 cm2 on one volar forearm (3) Unable to come to the infant's hospital for study measurements on one day when infant measurements are made (4) Unwilling to provide written informed consent for participation

-

Ages: 24 Weeks to 43 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants and parents of infants who are patients at Cincinnati Children's Hospital Medical Center Neonatal Intensive Care Units including premature and full-term infants
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Time for premature infants stratum corneum lipid composition to become indistinguishable from composition in healthy full term infants and in comparison to a contralateral site treated with sunflower oil | Until six months after discharge
  Stratum corneum ceramides, sphingoid bases, and free fatty acids in premature infants will be compared with those in full term infants and adults. The composition will be evaluated over six months for premature infants and full term infants and compared to those of adults. Lipid composition is determined from extracts of stratum corneum collected from the skin surface at designated skin sites on each leg. Analyses are conducted using supercritical fluid chromatography and tandem mass spectrometry and reported as total free fatty acids, cholesterol, total ceramides and total sphingoid bases normalized to total protein.

SECONDARY OUTCOMES:
Skin Surface Acidity | Until six months after discharge
  Skin surface acidity in premature infants will be compared to the lipid composition. The skin surface acidity and the lipid composition will be compared over time for premature and full term infants. An acidic skin surface is necessary for the effective functioning of enzymes in stratum formation and integrity and for bacterial homeostasis, skin colonization and inhibition of pathogenic bacteria. In very low birth weight infants, skin acidity varies with gestational age and is higher for a longer time compared with full term infants.

CONTACTS AND LOCATIONS:
Overall Officials: Marty O Visscher, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Cincinnati Childrens Hospital Medical Center Neonatal Intensive Care Unit, Cincinnati, Ohio
  - University Hospital Neonatal Intensive Care Unit, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No